CLINICAL TRIAL: NCT06588322
Title: Detection of Homologous Recombination Pathway Gene Mutations in Circulating Tumour DNA From BRCA-mutated Ovarian Cancer Patients Receiving First-line PARP Inhibitor Maintenance Therapy
Acronym: ATROVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24GENF01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with an epithelial ovarian cancer. (Other)
  Interventions: Other: Blood samples will be taken on several times (36 mL of blood taken at each time):

INTERVENTIONS:
Other: Blood samples will be taken on several times (36 mL of blood taken at each time): — * Inclusion visit (T0): prior to initiation of Olaparib treatment
  * Follow-up period (T1 to T8): every 3 months for a maximum of 24 months
  * End of study (Tx): on definitive cessation of Olaparib treatment for any reason (progression, toxicity or definitive cessation of treatment after 2 years).

SUMMARY:
This is an interventional (category 2), prospective, multicentric cohort study designed to demonstrate that the search, based on Circulating tumour DNA analysis, for a BRCA1/2 reversion mutation leading to restoration of its protein function enables early identification of disease progression in BRCA1/2 mutant patients treated as first-line maintenance with a PARP inhibitor (Olaparib alone or in combination with bevacizumab) for ovarian cancer.

For this study, a total of 9 blood samples will be taken from patients who will undergo a full 24-month treatment regimen.

Apart from the study procedure (blood sampling), all examinations carried out in this study, treatment with Olaparib (alone or combined with bevacizumab) and patient follow-up procedures will be carried out as part of routine care in accordance with the standard practices of each investigating site.

130 patients will take part in the study, and each patient will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an epithelial ovarian cancer, fallopian tube cancer or primitive of the peritoneum.
2. Patient with a BRCA 1 or 2 somatic and/or constitutional mutation previously confirmed and validated by an approved laboratory.
3. Patient due to start first-line maintenance treatment with Olaparib alone (PARP inhibitor) or in combination with bevacizumab.
4. Age ≥ 18 years at the time of signing the consent.
5. WHO ≤ 1.
6. Patient affiliated to a Social Security scheme in France.
7. Patient having signed informed consent prior to inclusion in the study and prior to any specific procedure for the study.

Exclusion Criteria:

1. Other cancer under treatment.
2. Olaparib treatment already initiated.
3. Indication for treatment with a PARP inhibitor other than Olaparib.
4. Any pathology contraindicating the sample collection procedures required by the study.
5. Any psychological, family, geographical or sociological condition that makes it impossible to comply with medical monitoring and/or the procedures laid down in the study protocol.
6. Subjects deprived of their liberty or under legal protection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
The rate of patients (in the population of patients with disease progression) with disease progression that was preceded by the detection of BRCA1/2 reversion mutation in circulating tumour DNA (i.e. Sensitivity). | 24 months for each patient
  Sensitivity is defined as the ratio of the number of disease progression events in which a reversion mutation was detected early to the number of disease progression events.

SECONDARY OUTCOMES:
The rate of patients with BRCA 1/2 reversion mutations at inclusion. | 24 months for each patient
  It is defined as the ratio of the number of patients with BRCA 1 / 2 reversion mutations at inclusion to the total number of patients.
Progression-free survival. | 24 months for each patient
  It is defined as the time between the date of inclusion and the date of progression or death from any cause. Patients alive without progression at the date of last news are censored.
The concordance between the type/location of the germline or somatic BRCA1/2 mutation and the BRCA1/2 reversion mutation will be presented in the form of a contingency table. | 24 months for each patient
The rates of patients with mutations in the other genes of the HR pathway at inclusion and at relapse. | 24 months for each patient
  It will be defined respectively by the ratio of the number of patients with reversion mutations at inclusion to the total number of patients and by the ratio of the number of patients with reversion mutations at relapse to the total number of patients with relapse.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Site Angers, Angers
  - Institut Bergonie, Bordeaux
  - Chu de Limoges, Limoges
  - Chu de Nimes, Nîmes
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Site Saint-Herblain, Saint-Herblain
  - IUCT-O, Toulouse